CLINICAL TRIAL: NCT02843074
Title: Phase 2 Study Assessing Feasibility and Tolerance of the Combination of Elotuzumab, Lenalidomide and Dexamethasone in Induction, Consolidation and Maintenance Treatment of Transplant-Eligible Patients Newly Diagnosed With Multiple Myeloma
Brief Title: Elotuzumab, Lenalidomide and Dexamethasone in Treatment of Transplant-Eligible Newly Diagnosed Multiple Myeloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MM61
Record Dates: First submitted 2016-07-20; First posted 2016-07-25 (Estimated); Results first posted 2022-10-17 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
Keywords: B-cell tumors; autologous stem cell transplantation; blood cancers
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms | interventions — elotuzumab; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ERd Therapy (Experimental): INDUCTION:
  Cycles 1-2: elotuzumab 10mg/kg IV days 1, 8, 15, 22; lenalidomide (len) 25mg orally (PO), once daily (QD) on days 1-21; dexamethasone (dex) 28 mg PO (3-24 hrs before elotuzumab IV) and 8mg IV (45-90 minutes before elotuzumab) days 1, 8, 15, 22.
  Cycles 3-4: elotuzumab 10mg/kg IV days 1 and 15; len 25mg PO QD days 1-21; dex 8mg PO (3-24 hrs before elotuzumab IV) and 8mg IV (45-90 minutes before elotuzumab) days 1 and 15; dex 40mg PO days 8 and 22.
  CONSOLIDATION:
  Four 28-day cycles: elotuzumab 10mg/kg IV days 1 and 15; len 15mg PO QD days 1-21; dex 28mg PO (3-24 hrs before elotuzumab) and 8mg IV (45-90 minutes before elotuzumab) days 1 and 15; dex 40mg PO days 8 and 22.
  MAINTENANCE:
  After completing consolidation therapy patients without progressive disease will receive, for up to 24 months, 28-day cycles of elotuzumab 20mg/kg IV day 1; len 10mg +/- 5mg PO QD days 1-21; dex 28mg PO (3-24 hrs before elotuzumab) and 8mg IV (45-90 minutes prior to elotuzumab) day 1.
  Interventions: Drug: elotuzumab; Drug: Lenalidomide; Drug: Dexamethasone; Procedure: autologous stem cell transplantation

INTERVENTIONS:
Drug: elotuzumab — Given intravenously (IV)
  Other Names: Empliciti
Drug: Lenalidomide — Given by IV
  Other Names: Revlimid
Drug: Dexamethasone — Given orally (PO) or by IV
  Other Names: Decadron
Procedure: autologous stem cell transplantation
  Other Names: ASCT

SUMMARY:
This is a phase 2, single arm, open-label, multicenter study to evaluate the feasibility and tolerance of the combination of elotuzumab, lenalidomide, and dexamethasone in the induction, consolidation, and maintenance treatment of transplant eligible, newly diagnosed multiple myeloma patients.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the feasibility of using the combination of elotuzumab, lenalidomide, and dexamethasone (ERd) as induction therapy and the ability of the combination to facilitate the start of autologous stem cell transplantation (ASCT) in transplant-eligible patients newly diagnosed with multiple myeloma. In addition to induction, the efficacy, safety, and tolerability of ERd as consolidation and maintenance therapy in these patients will be observed.

Eligible patients will undergo four 28-day cycles of an induction regimen of elotuzumab, lenalidomide, and dexamethasone. Following completion of 4 cycles of induction therapy, all patients will undergo standard mobilization, collection of stem cells, and then ASCT using a melphalan conditioning regimen as per institutional guidelines.

Toxicity evaluation will be interrupted during the stem cell procedure and will resume with the onset of consolidation. Adverse events will be collected, however, from the end of induction up to mobilization.

Consolidation therapy will begin 70 to 120 days following ASCT and will consist of four 28-day cycles of elotuzumab, lenalidomide, and dexamethasone. All patients that do not experience progressive disease will begin maintenance therapy of elotuzumab, lenalidomide, and dexamethasone. The duration of maintenance will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed myeloma requiring systemic chemotherapy as per International Myeloma Working Group (IMWG) uniform criteria and Diagnostic Criteria and Staging for Multiple Myeloma

  * Ideally, no prior therapy, or
  * No more than 1 cycle of therapy for emergent control of disease prior to enrolling on study, including prior treatment of hypercalcemia, spinal cord compression, or active and/or aggressively progressing myeloma with corticosteroids or lenalidomide or bortezomib-based regimens (treatment dose should not exceed the equivalent of 160 mg of dexamethasone in a 4 week period, or not more than 1 cycle)
  * Bisphosphonates are permitted
* Eligible and plan to undergo ASCT in first remission
* Measurable disease, prior to initial treatment as indicated by one or more of the following:

  * Serum M-protein ≥1.0 g/dL
  * Urine M-protein ≥200 mg/24 hours
  * Serum free light chain assay: involved free light chain level ≥10 mg/dL (≥100 mg/L) provided the serum free light chain ratio is abnormal.
* Ability to take aspirin or other venous thromboembolism (VTE) anticoagulant therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 thru 2
* Adequate hematologic, renal, and liver function.
* All study participants must be registered into the mandatory Revlimid REMS® program and must be willing and able to comply with the requirements of that program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Male patients with female partners of childbearing potential and female patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 28 days following last dose of study drugs. Male patients must also refrain from donating semen or sperm during their participation in the study.
* Willingness and ability to comply with study and follow-up procedures.
* Ability to understand the nature of this study and give written informed consent.

Exclusion Criteria:

* Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes (POEMS) syndrome
* Plasma cell leukemia
* Waldenström's macroglobulinemia or IgM myeloma
* Presence of other active cancers, or history of treatment for invasive cancer ≤5 years. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with a history of non-melanoma skin cancer.
* Radiotherapy to multiple sites or immunotherapy within 4 weeks before start of protocol treatment (localized radiotherapy to a single site at least 1 week before start is permissible)
* Major surgical procedures ≤28 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement.
* Acute active infection requiring systemic antibiotics, antivirals, or antifungals within 2 weeks prior to first dose of study treatment
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea Grade ≥2, and malabsorption syndrome)
* Any of the following cardiac diseases currently or within the last 6 months:

  * Left ventricular ejection fraction (LVEF) <40% as determined by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan
  * Unstable angina pectoris
  * Congestive heart failure (New York Heart Association ≥ Grade 2
  * Acute myocardial infarction
  * Conduction abnormality not controlled with pacemaker or medication
  * Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
  * Valvular disease with significant compromise in cardiac function
* Known seropositive for or active viral infection with human immunodeficiency virus or hepatitis A, B, or C virus. Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Any clinically significant medical disease or condition that, in the treating Investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent
* Pregnant or lactating females
* Contraindication to any of the required concomitant drugs, including dexamethasone, H1 and H2 blockers, and acetaminophen, or if patient has a history of prior thrombotic disease, warfarin or low molecular weight heparin
* No health coverage, or if the copay for lenalidomide is not acceptable to the patient.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Berdeja, MD, Study Chair — SCRI Development Innovations, LLC
Locations (6):
- United States (6):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - HCA Midwest Health/Research Medical Center, Kansas City, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew consent before the study treatment assignment.
Groups:
- ERd Therapy: INDUCTION:
  Cycles 1-2: elotuzumab 10mg/kg IV days 1, 8, 15, 22; lenalidomide (len) 25mg orally (PO), once daily (QD) on days 1-21; dexamethasone (dex) 28 mg PO (3-24 hrs before elotuzumab IV) and 8mg IV (45-90 minutes before elotuzumab) days 1, 8, 15, 22.
  Cycles 3-4: elotuzumab 10mg/kg IV days 1 and 15; len 25mg PO QD days 1-21; dex 8mg PO (3-24 hrs before elotuzumab IV) and 8mg IV (45-90 minutes before elotuzumab) days 1 and 15; dex 40mg PO days 8 and 22.
  CONSOLIDATION:
  Four 28-day cycles: elotuzumab 10mg/kg IV days 1 and 15; len 15mg PO QD days 1-21; dex 28mg PO (3-24 hrs before elotuzumab) and 8mg IV (45-90 minutes before elotuzumab) days 1 and 15; dex 40mg PO days 8 and 22.
  MAINTENANCE:
  After completing consolidation therapy patients without progressive disease will receive, for up to 24 months, 28-day cycles of elotuzumab 20mg/kg IV day 1; len 10mg +/- 5mg PO QD days 1-21; dex 28mg PO (3-24 hrs before elotuzumab) and 8mg IV (45-90 minutes prior to elotuzumab) day 1.
  elotuzumab: Given intravenously (IV)
  Lenalidomide: Given by IV
  Dexamethasone: Given orally (PO) or by IV
  autologous stem cell transplantation
Period: Overall Study
Arm/Group | ERd Therapy
Started | 52
Completed | 35
Not Completed | 17
Not completed — Withdrawal by Subject | 5
Not completed — Progressive disease | 1
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Death | 9

BASELINE CHARACTERISTICS:
Arm/Group | ERd Therapy
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Induction Feasibility Rate (IFR)
Description: Defined as the percentage of patients who successfully complete four 28-day cycles of induction therapy with elotuzumab, lenalidomide and dexamethasone (ERd) and start autologous stem cell transplantation (ASCT).
Time Frame: approximately 22 weeks (16 weeks of treatment and 6 weeks allowance for planning and scheduling mobilization and ASCT).
Population: Four participants who completed four 28-day cycles of induction therapy refused transplantation (ASCT). These 4 participants were excluded from the IFR analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ERd Therapy
Number analyzed (Participants) | 48
Participants | 33

2. Secondary Outcome: Complete Response Rate (CRR) for Complete Time on Study
Description: Defined as the percentage of patients who achieve a complete response (CR) or near complete response (nCR) to treatment at each stage of the study (induction, ASCT, consolidation, end of study) per International Myeloma Working Group (IMWG) and European Group for Blood and Marrow Transplantation (EBMT) criteria.CR=bone marrow contains ≤5% plasma cells; negative immunofixation on serum and urine; disappearance of soft tissue plasmacytomas. nCR = the absence of myeloma protein on electrophoresis, with positive immunofixation, stable bone disease, and a normal serum calcium concentration. Patient must have completed at least 1 cycle to be included in analysis.
Time Frame: every 4 weeks until end of treatment visit, and every 3 months thereafter up to 3 years
Population: Participants who completed at least one cycle of treatment were included in the analysis. One participant didn't complete cycle 1 due to adverse events; therefore, excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ERd Therapy
Number analyzed (Participants) | 51
Participants | 25

3. Secondary Outcome: Overall Response Rate (ORR) for Complete Time on Study
Description: Defined as percentage of patients receiving at least 1 cycle with confirmed complete response, very good partial response, or partial response (CR, VGPR, or PR) to treatment at each stage of the study (induction, ASCT, consolidation, end of study) per IMWG and EBMT criteria. CR=bone marrow contains ≤5% plasma cells; negative fixation on serum and urine; the disappearance of soft tissue plasmacytomas. VGPR=serum and urine M-protein detectable by immunofixation but not by electrophoresis or ≥90% reduction from baseline serum and urine M-protein level <100mg for 24h and In case of presence of soft tissue plasmacytoma(s) at baseline, the disappearance of any soft tissue plasmacytomas. PR=≥50% reduction from baseline in serum M-protein and ≥90% reduction from baseline in 24h urinary M-protein or urine M-protein <200 mg/24 hours and In case of presence of soft tissue plasmacytoma(s) at baseline, a reduction in the sum of products of the two longest perpendicular diameters (SPD) by >50%.
Time Frame: every 4 weeks until end of treatment visit, and every 3 months thereafter up to 3 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ERd Therapy
Number analyzed (Participants) | 51
Participants | 47

4. Secondary Outcome: Progression-free Survival (PFS)
Description: The time from start of induction treatment to documented progressive disease (PD) or death from any cause up to 3 years post first study treatment. PD is defined as an increase of ≥ 25% from the nadir in at least one of the following criteria: serum M-protein (absolute increase must be ≥0.5 g/dL); urine M-protein (absolute increase must be ≥200 mg/24h) ; only in patients with non-measurable serum and urine M-protein levels: difference in involved and uninvolved FLC levels (absolute increase must be >10 mg/dL); only in patients with non-measurable serum and urine M-protein levels and non-measurable disease by FLC levels, bone marrow plasma cell % (absolute % must be ≥10%) OR Definite development of new bone lesions or soft tissue plasmacytomas OR definite increase in the size of existing bone lesions or soft tissue plasmacytomas OR Development of hypercalcemia (corrected serum Ca >11.5mg/dL) for patients without hypercalcemia at baseline. Must have completed 1 cycle to be included.
Time Frame: every 4 weeks until end of treatment visit, and every 3 months thereafter up to 3 years
Population: as for outcome 2
Measure: Median (99% Confidence Interval); unit: months
Arm/Group | ERd Therapy
Number analyzed (Participants) | 51
months | 29.7002 [20.53 to NA] — The upper limit of the 99% CI is not estimable by Kaplan-Meier method based on the data and events collected.

5. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from start of induction treatment to 3 years post first study treatment or death from any cause, whichever comes first. Patient must have completed at least 1 cycle to be included in analysis.
Time Frame: every 4 weeks until end of treatment visit, and up to 3 years thereafter
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | ERd Therapy
Number analyzed (Participants) | 51
months | NA [NA to NA] — Since only a few patients died, the median survival was not estimable by Kaplan-Meier method nor the 90% confidence interval.

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events as a Measure of Safety
Description: Safety data and abnormal lab values and abnormal vital signs were collected and assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE V4.03).
Time Frame: weekly for 8 weeks, then every 2 weeks till the start of mobilization for Induction and 70-120 days post-ASCT, every 2 weeks during 16 weeks of Consolidation, and monthly for 24 months of Maintenance, up to 30 days after last dose of study drugs.
Population: All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | ERd Therapy
Number analyzed (Participants) | 52
Participants | 52

7. Secondary Outcome: Consolidation Feasibility Rate (CFR)
Description: defined as the percentage of patients starting induction treatment with ERd successfully completing treatment to end of consolidation
Time Frame: approximately 55 weeks (16 weeks of induction treatment, 6 weeks allowance for planning and scheduling mobilization and ASCT, 17 weeks pause in treatment after ASCT, 16 weeks of consolidation treatment).
Population: All patients starting induction treatment
Measure: Count of Participants; unit: Participants
Arm/Group | ERd Therapy
Number analyzed (Participants) | 52
Participants | 34

8. Secondary Outcome: Maintenance Feasibility Rate (MFR)
Description: defined as the percentage of patients starting induction treatment with ERd successfully completing treatment to end of maintenance
Time Frame: approximately 159 weeks (16 weeks of induction treatment, 6 weeks allowance for planning and scheduling mobilization and ASCT, 17 weeks pause in treatment after ASCT, 16 weeks of consolidation treatment, 104 weeks/2 years of maintenance treatment)
Population: All patients starting induction treatment
Measure: Count of Participants; unit: Participants
Arm/Group | ERd Therapy
Number analyzed (Participants) | 52
Participants | 19

ADVERSE EVENTS:
Time Frame: weekly for 8 weeks, then every 2 weeks till the start of mobilization for Induction treatment and 70-120 days post-ASCT, every 2 weeks during 16 weeks of Consolidation treatment, and monthly for 24 months of Maintenance treatment up to 30 days after last dose of study drugs.
Description: Assessments will be made through analysis of the reported incidence of treatment-emergent Serious Adverse Events (SAEs) and non-serious adverse events (AEs).
Arm/Group | ERd Therapy
All-Cause Mortality (participants affected / at risk) | 9/52
Serious Adverse Events (participants affected / at risk) | 20/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERd Therapy (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (2)
Cardiac perforation (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERd Therapy (N=52)
Anaemia (Blood and lymphatic system disorders) | 10 (29)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 9 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (15)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Deafness (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 7 (7)
Ectropion (Eye disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (3)
Visual impairment (Eye disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 2 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (6)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 20 (31)
Diarrhoea (Gastrointestinal disorders) | 25 (39)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (8)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 22 (31)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Poor dental condition (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (15)
Asthenia (General disorders) | 7 (7)
Chest discomfort (General disorders) | 1 (1)
Chills (General disorders) | 10 (12)
Fatigue (General disorders) | 31 (48)
Feeling abnormal (General disorders) | 1 (1)
Feeling cold (General disorders) | 1 (1)
Feeling jittery (General disorders) | 1 (1)
Influenza like illness (General disorders) | 6 (12)
Infusion site bruising (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 4 (5)
Non-cardiac chest pain (General disorders) | 2 (2)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 10 (10)
Pain (General disorders) | 6 (6)
Peripheral swelling (General disorders) | 6 (7)
Pyrexia (General disorders) | 18 (33)
Temperature intolerance (General disorders) | 1 (1)
Unevaluable event (General disorders) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 4 (4)
Bronchitis (Infections and infestations) | 4 (4)
Candida infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (9)
Rhinitis (Infections and infestations) | 3 (4)
Rhinovirus infection (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 4 (6)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (12)
Urinary tract infection (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural erythema (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (8)
Blood bilirubin increased (Investigations) | 1 (2)
Blood creatinine increased (Investigations) | 3 (3)
Blood glucose increased (Investigations) | 1 (2)
Blood immunoglobulin G decreased (Investigations) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 2 (2)
Blood potassium decreased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 2 (2)
Breath sounds abnormal (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Immunoglobulins decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (6)
Platelet count decreased (Investigations) | 2 (2)
Weight decreased (Investigations) | 4 (6)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 17 (19)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (11)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (8)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (19)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (17)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 (23)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (2)
Disturbance in attention (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 6 (7)
Dizziness postural (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 3 (3)
Dysgraphia (Nervous system disorders) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 11 (15)
Hyperaesthesia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 4 (4)
Hypogeusia (Nervous system disorders) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 13 (21)
Paraesthesia (Nervous system disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Restless legs syndrome (Nervous system disorders) | 1 (2)
Sensory disturbance (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 4 (5)
Taste disorder (Nervous system disorders) | 3 (4)
Tremor (Nervous system disorders) | 4 (5)
Affect lability (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 8 (8)
Confusional state (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 6 (7)
Disorientation (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 16 (18)
Irritability (Psychiatric disorders) | 2 (2)
Libido decreased (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (21)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (15)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 7 (7)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 12 (17)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Aortic dilatation (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Flushing (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 1 (4)
Pallor (Vascular disorders) | 1 (2)
Phlebitis (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT02843074/Prot_SAP_000.pdf